CLINICAL TRIAL: NCT00726609
Title: Post-marketing Surveillance (PMS) Management of Invasive Mycosis With Posaconazole
Brief Title: Post-marketing Surveillance Study of Invasive Mycosis With Posaconazole (Study P04641)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04641
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2009-09-22 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Posaconazole (assigned by physician in normal practice): * Treatment of invasive fungal infection.
  * Prophylaxis of invasive fungal infection.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — The usual dose of NOXAFIL® is 400 mg twice daily (10 mL) at meals or with 240 mL of a food supplement. For patients unable to take meals or food supplements, NOXAFIL® is administered at a dose of 200 mg (5 mL) four times daily.
  Other Names: SCH 56592; NOXAFIL®

SUMMARY:
The purpose of this postmarketing surveillance study is to collect an extensive body of data in a large patient population in every day life to investigate the safety and efficacy of NOXAFIL® (posaconazole) in the treatment of invasive fungal disease.

DETAILED DESCRIPTION:
Data regarding demographics, underlying disease, prior fungal infection, prior antifungal medication, invasive fungal infection signs & symptoms, concomitant medication, posaconazole use, tolerability, safety and therapy outcome will be collected on abstracted electronic Case Report Forms.

This surveillance study was originally limited to subjects receiving posaconazole as salvage antifungal therapy as indicated. A subgroup of subjects at risk for invasive fungal infection was included for prophylactic treatment following the enlargement of the marketing authorization for NOXAFIL® (posaconazole) during the course of the study. These participants only contributed data for the assessment of safety.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects with:

* Invasive aspergillosis refractory to, or intolerant of, amphotericin B or itraconazole,
* Fusariosis refractory to, or intolerant of, amphotericin B,
* Chromoblastomycosis and mycetoma refractory to, or intolerant of, itraconazole,
* Coccidiomycosis refractory to, or intolerant of, amphotericin B, itraconazole or fluconazole.
* Subjects receiving remission-induction chemotherapy for acute myelogenous leukemia (AML) or myelodysplastic syndromes (MDS) expected to result in prolonged neutropenia and who are at high risk for developing invasive fungal infections.
* Hematopoietic stem-cell transplant (HSCT) recipients who are undergoing high-dose immunosuppressive therapy for Graft-versus-host disease and who are at high risk for developing invasive fungal infections.

Exclusion Criteria:

* Comedication of the participant with ergotamine, dihydroergotamine, terfenadine, astemizole, cisapride, pimozide, halofantrine, or chinidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with invasive fungal infection refractory to first-line treatment or unable to tolerate it were selected at hospitals in Germany.
  Following the enlargement of the marketing authorization for posaconazole, subjects at risk for invasive fungal infection were also enrolled.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posaconazole (Assigned by Physician in Normal Practice)
Started | 214
Completed | 116 (For 26 participants in the Missing category, it is unknown if they completed the study.)
Not Completed | 98
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 25
Not completed — Other | 16
Not completed — Missing | 42
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole (Assigned by Physician in Normal Practice)
Number analyzed (Participants) | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 135
Region of Enrollment [Number; unit: participants]
  Germany | 214

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Drug Reactions.
Description: The severity of an Adverse Drug Reaction is determined on the basis of the following definitions:
  Mild: The abnormality, symptom or event is noticed but well tolerated.
  Moderate: Symptoms impair normal activities and may require intervention.
  Severe: Clinical status is significantly impaired, normal activity is no longer possible, intervention is required.
Time Frame: Before starting treatment with posaconazole, during treatment, and until 100 days after treatment.
Measure: Number; unit: Participants
Arm/Group | Posaconazole (Assigned by Physician in Normal Practice)
Number analyzed (Participants) | 214
Participants
  All | 52
  Mild | 30
  Moderate | 21
  Severe | 1

ADVERSE EVENTS:
Arm/Group | Posaconazole (Assigned by Physician in Normal Practice)
Serious Adverse Events (participants affected / at risk) | 33/214
Other Adverse Events (participants affected / at risk) | 49/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (Assigned by Physician in Normal Practice) (N=214)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1)
CYSTIC LYMPHANGIOMA (Congenital, familial and genetic disorders) | 1 (1)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
DEATH (General disorders) | 2 (2)
DISEASE PROGRESSION (General disorders) | 2 (2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1)
INJECTION SITE THROMBOSIS (General disorders) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 2 (3)
PYREXIA (General disorders) | 1 (2)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1)
ACUTE GRAFT VERSUS HOST DISEASE (Immune system disorders) | 1 (1)
ACUTE GRAFT VERSUS HOST DISEASE IN INTESTINE (Immune system disorders) | 1 (1)
ACUTE GRAFT VERSUS HOST DISEASE IN LIVER (Immune system disorders) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 1 (1)
ABSCESS SWEAT GLAND (Infections and infestations) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 4 (4)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 2 (3)
INFECTION (Infections and infestations) | 2 (2)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1)
OTITIS MEDIA BACTERIAL (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
SKIN INFECTION (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 6 (10)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 2 (2)
UROSEPSIS (Infections and infestations) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
BLOOD CULTURE POSITIVE (Investigations) | 1 (4)
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 2 (2)
RENAL FUNCTION TEST ABNORMAL (Investigations) | 2 (2)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 1 (1)
ENCEPHALITIS (Nervous system disorders) | 1 (1)
TOXIC NEUROPATHY (Nervous system disorders) | 1 (1)
TRANSIENT PSYCHOSIS (Psychiatric disorders) | 1 (1)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (Assigned by Physician in Normal Practice) (N=214)
DIARRHOEA (Gastrointestinal disorders) | 19 (19)
NAUSEA (Gastrointestinal disorders) | 12 (18)
PYREXIA (General disorders) | 27 (34)
C-REACTIVE PROTEIN INCREASED (Investigations) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No